CLINICAL TRIAL: NCT06108505
Title: A Prospective, Multicentre, Randomised Clinical Study Evaluating the Effectiveness of Lacticaseibacillus Wild Type Strain on Lowering Blood Cholesterol Levels
Brief Title: A Clinical Study on the Effectiveness of a Lacticaseibacillus Strain on Blood Cholesterol Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Yiannis Kourkoutas, Laboratory of Applied Microbiology & Biotechnology, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLASSIC study
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cholesterol Levels

STUDY DESIGN:
Intervention Model Description: A 1:1 randomization will be used in the study to allocate subjects into two groups. A group will receive the strain of Lacticaseibacillus with oats and the other group will receive only plain oats.
Who Masked: Participant, Investigator
Masking Description: Neither participant nor site investigator is aware for the product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacticaseibacillus with oats (Experimental): This group of subjects receives the Lacticaseibacillus with oats.
  Interventions: Other: Lacticaseibacillus with oats
- Plain oats (Placebo Comparator): This group of subjects receives plain oats.
  Interventions: Other: Plain oats

INTERVENTIONS:
Other: Lacticaseibacillus with oats — Subjects will receive 7.5 gr of oats containing Lacticaseibacillus
  Arms: Lacticaseibacillus with oats
Other: Plain oats — Subjects will receive 7.5 gr of plain oats
  Arms: Plain oats

SUMMARY:
This is a 12-week prospective, multicentre, randomised Phase 4 study to evaluate the effect of a wild type strain of Lacticaseibacillus in cholesterol of blood levels.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effect of a wild type strain of Lacticaseibacillus as an incorporated ingredient of oat powder in the improvement of low density lipoprotein levels. In the study will participate two groups of subjects, one group with receive the strain with oats for 2.5 months and the other a group of subjects will receive plain oats. During the study, the subjects will receive only the product of the study and no other intervention will be performed except the standard clinical practice. The subjects will perform 4 visits and their eligibility will be evaluated at the baseline visit by performing routine clinical and laboratory examinations. The subjects who will consent to participate in the study will be randomised 1:1 into one of the study arms (Lacticaseibacillus and oats vs. oats). At each follow-up visit, the standard clinical and laboratory tests for dyslipidemia will be performed at the hospital.

Following a treatment period of 10 weeks, a 2-week washout observational period will take place where subjects will not receive any product.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants of either sex with ages between 18 and 70 years (limits included).
2. Participants with serum LDL-C ≥116 mg/dl.
3. Body Mass Index (BMI) between 18.5 and 35 kg/m2 (limits excluded).

Exclusion Criteria:

1. Subjects who systematically receive any other lipid-lowering non-medicinal product, supplement or functional food such as ACTIMEL, ACTIVIA, oat beta-glucan, pharmaceutical garlic, or stopped less than 1 month prior to study inclusion.
2. Participants that have been under lipid-lowering drug treatment (e.g. statins, fibrates, etc.) or any other medication that has a significant effect on LDL-c within the last 2 months prior to study inclusion.
3. Lactating females or those that are planning pregnancy within 6 months from the start of the study.
4. Participants with a history of ischemic cardiovascular events, alcohol abuse, or suffering from a severe chronic disease (e.g. cancer, diabetes, chronic advanced kidney disease, thyroid disorders, hepatic disorders, cancer, familial hypercholesterolemia or immunosuppression) that would potentially affect the outcomes of the study.
5. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
6. Subjects with a known intolerance or allergy to any ingredient of the administered products.
7. Participants who are planning on making significant changes in their diet, lifestyle, and physical activity during the duration of the study, i.e. participants that are currently on weight-reducing diets.
8. Participants who are receiving any interventional procedure or are currently included in a clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
LDL-c levels up to 10 weeks | At 10 weeks after treatment initiation
  Change in LDL-c levels from baseline at 10 weeks

SECONDARY OUTCOMES:
LDL-c levels up to 12 weeks | At 6 and 12 weeks after treatment initiation
  Change in LDL-c levels from baseline at 6 and 12 weeks
HDL-c, total cholesterol, and TG levels measurement | At 6, 10 and 12 weeks after treatment initiation
  Change in HDL-c, total cholesterol, and TG levels from baseline at 6, 10, and 12 weeks
Changes in SCORE 2 levels | At 10 weeks after treatment initiation
  Change in SCORE2 risk level from baseline at 10 weeks
Subjects adherence to study | Up to 10 weeks
  The percentage of participants that are adherent to receiving the study product, defined as receiving ≥80% off suggested doses at 10 weeks
Serious adverse events evaluation | Up to 12 weeks after treatment initiation
  The number, type, severity, and seriousness of adverse events related to the study product

OTHER OUTCOMES:
Changes in VAS scale | At 6, 10 and 12 weeks
  Change in 11-point Visual Activity Score (VAS) from baseline on the overall satisfaction with bowel symptoms and Bristol Stool scale at 6, 10, and 12 weeks.
Changes in serum levels | At 6, 10 and 12 weeks
  Change in the serum levels, compared to baseline, of glucose, creatinine, urea, AST, ALT, γGT, ALP, LDH, hsCRP, and Lp(a), ΑpoA1, ApoB, Homocysteine, vitD as optional, where available, at 6, 10, and 12 weeks
Changes in LDL-c, HDL-c, total cholesterol, and TG | Up to 12 weeks
  Change in LDL-c, HDL-c, total cholesterol, and TG at each visit compared to levels within 3 months before study inclusion, where available, and for patients who did not receive any therapeutic or lifestyle interventions during that time

CONTACTS AND LOCATIONS:
Overall Officials: Yiannis Kourkoutas, Study Director — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, East Macedonia and Thrace, Greece

IPD SHARING:
Plan to Share IPD: No
Only aggregates results can be available for GDPR reasons